CLINICAL TRIAL: NCT06372860
Title: Diabetes Prevention Program Feasibility Study of Breastfeeding - Electronic Monitoring of Mom's Schedule 2.0
Brief Title: DPP Feasibility Study of Breastfeeding - eMOMS 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Ascension Health (Industry); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lisette Jacobson, Associate Professor, Population Health, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RKS2018350; 3P20GM144269-02S2 (NIH)
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Overweight or Obesity; Pregnancy
Keywords: diabetes prevention; breastfeeding; lactation support; prediabetes
MeSH Terms: conditions — Overweight; Obesity; Breast Feeding; Prediabetic State | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP + Breastfeeding (Tx1) (Active Comparator): Patients randomized to Tx1 will receive education in the Diabetes Prevention Program (DPP) and intensive breastfeeding education and support. Ante- and postpartum education includes access to the mHealth app and individualized 1-on-1 health coaching. Phase I is delivered antepartum and includes: four (4) 1-hour DPP-based educational sessions and six (6) 20-minute educational videos on lactation. Phase II is delivered postpartum and includes: in-hospital lactation support and two (2) 1-hour DPP-based educational sessions. Participants will continue to receive individualized 1-on-1 health coaching through 3 months postpartum.
  Interventions: Behavioral: Diabetes Prevention Program; Behavioral: Breastfeeding; Behavioral: Usual Care
- Usual Care (Placebo Comparator): Usual care is described as obstetrical care that pregnant women with normal BMI receive and that is provided by their provider. There will not be any antepartum education or 1-on-1 health coaching. Postpartum education will only include usual care in-hospital lactation support. There will not be any other education nor 1-on-1 support.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — The intervention will be administered by professionally trained, certified health coaches. Phase I consists of four 1-hour DPP-based sessions to be completed during pregnancy. Each session will be pre-recorded and archived on a secure, private mHealth application. Participants will be asked to complete each session on their own time. A health coach will follow up weekly via phone to check on progress and will work with the participant 1-on-1, if needed. Phase I will be completed by week 36 of pregnancy. Prior to delivery, participants are invited to a virtual focus group about their experiences.
  Phase II consists of two 1-hour DPP-based sessions to be completed after delivery. Each session will be pre-recorded and archived on the same mHealth application. Participants will begin Phase II within 1 week of delivery with the same health coach. Phase II will be completed by week 12 postpartum. Upon completion, participants are invited to a virtual focus group about their experiences.
  Arms: DPP + Breastfeeding (Tx1)
Behavioral: Breastfeeding — Phase I also consists of six (6) breastfeeding videos that are pre-recorded into 15-20 minute sessions and will be available on the mHealth application. Participants will have access to the first 2 sessions by week 28 of pregnancy and need to complete the remaining 4 sessions by week 36 of pregnancy. Each session is taught by an International Board Certified Lactation Consultant (IBCLC).
  Participants will receive 1-on-1 lactation support by the same DPP health coach. The health coach is a professionally trained Certified Breastfeeding Specialist (CBS). She will assist participants with any questions related to lactation. If the health coach is unable to help with a specific issue, she will contact the IBCLC-of-record, who will provide assistance to the health coach only. If the health coach or IBCLC deems additional care necessary, the participant will be referred to their primary care physician. The IBCLC will not have direct contact with the study participants.
  Arms: DPP + Breastfeeding (Tx1)
Behavioral: Usual Care — Participants will receive regular prenatal care provided by their physician. At delivery, all participants will receive some type of lactation support in the hospital.

SUMMARY:
The purpose of this study is to investigate the impact of a comprehensive intervention that combines breastfeeding support with a diabetes prevention-based program (DPP) on postpartum weight retention and lactation duration among women with pre-pregnancy overweight or obesity. This intervention, named eMOMS, is delivered by a certified health coach via a mobile health (mHealth) application.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to determine the feasibility and efficacy of a combined breastfeeding, diabetes prevention-based program (DPP) in a cohort of overweight or obese women to be followed during pregnancy through 3 months postpartum. The trial will have two study arms: DPP + breastfeeding (Tx1) and Usual Care (Tx2).

Aim 1: Quantify interest in use of the DPP-lactation mobile health (mHealth) application among target population. To accomplish this, we will: (1) measure research engagement including rates of screening, recruitment, and retention among users, especially rural and racially/ethnically diverse women; (2) assess barriers/facilitators to enrollment/retention through surveys and semi-structured in-depth interviews or focus groups; and (3) evaluate intervention uptake, delivery, and adherence via tracking/measuring use of the mHealth app.

Aim 2: Measure weight loss and duration of lactation through 3 months postpartum among target population. To accomplish this, we will measure pre-pregnancy weight, weight at study entry, weight immediately prior to and after delivery, and weight at specific postpartum time points. Lactation and infant feeding practices will be measured at similar postpartum time points.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* In second trimester or early third trimester
* BMI >/= 25 and < 35
* At least 18 years old or older
* Able to read and understand English
* Able to learn and use a video platform

Exclusion Criteria:

* Complications related to pregnancy that require emergency care
* Thyroid disease
* Multiple gestation
* Substance abuse within last 3 years
* Assisted reproductive technology (ART)-related pregnancy
* Current smoker
* Prior bariatric surgery
* In weight-loss program within 3 months of conception
* BMI >/= 35
* Unable to attend intervention/ follow-up visits
* Unwilling to self-monitor data collection
* Unable to complete intervention
* Presence of any condition that limits walking
* Presence of any condition that limits following diet recommendations
* Pregnancies complicated with fetuses diagnosed with lethal malformations/conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant must be a pregnant female.
Enrollment: 43 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Maternal weight | At baseline; at week 30, 32, and 34 of pregnancy; and at day 3, 10, week 3, 6, month 2 and month 3 postpartum.
  The study team will measure maternal weight to calculate maternal BMI and to allow for meaningful comparisons of weight change among study arms.
Maternal body mass index (BMI) | At baseline; at week 30, 32, and 34 of pregnancy; and at day 3, 10, week 3, 6, month 2 and month 3 postpartum.
  Body mass index (BMI) is a measure of body fat based on height and weight. The study team will measure BMI and to allow for meaningful comparisons of weight change among study arms.
Initiation of Lactation | At delivery.
  The study team will assess whether (yes/no) lactation was initiated at birth.
Duration of Lactation | At delivery, discharge, at day 7, week 3, 6, month 1, 2, and 3 postpartum.
  The study team will measure duration of maternal ability to breastfeed at specific timepoints.
Type of Infant Feeding | At delivery, discharge, at day 7, week 3, 6, month 1, 2, and 3 postpartum.
  The study team will measure "exclusive" lactation (human milk only) versus "any" lactation (predominant human milk with formula or solid food supplementation) at specific timepoints.

SECONDARY OUTCOMES:
Recruitment Rate | This will occur between day 1 of first participant enrollment through study completion, roughly 1-1.5 years.
  To assess recruitment rate, the study team will track the percent (%) of potential participants contacted versus the percent (%) of participants enrolled in the study.
Retention Rate | This will occur between day 1 of first participant enrollment through study completion, roughly 1-1.5 years.
  To assess retention rate, the study team will track the percent (%) of participants who complete the intervention.
Research Engagement | After week 36 of pregnancy but prior to delivery, and after month 3 postpartum.
  Participants who complete each phase of the program will be invited to participate in focus groups to discuss program experiences.
Mobile Application Usage | This will occur between day 1 of first participant enrollment through study completion, roughly 1-1.5 years.
  To assess intervention uptake, the study team will track the amount of time spent on each session on the mobile app.
Health Coach Interaction | This will occur between day 1 of first participant enrollment through study completion, roughly 1-1.5 years.
  To assess intervention uptake, the study team will track the amount of time spent with the health coach.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Jacobson, PhD, MPA, MA, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Via Christi Maternal Fetal Medicine Clinic, Wichita, Kansas, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT06372860/Prot_SAP_000.pdf